CLINICAL TRIAL: NCT06827288
Title: Adaptive Interventions for Emergency Department Patients With Opioid Use Disorder
Acronym: ADAPT-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Arrowhead Regional Medical Center (Other); Alameda Health System (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Katherine Watkins, Katherine Watkins, MD, RAND
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-N0631
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Solar System; Breath Holding

STUDY DESIGN:
Intervention Model Description: A two-stage Sequential Multiple Assignment Randomized Trial (SMART).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SUN with no follow up (Active Comparator): In Arm A, participants are randomized to receive SUN-assisted treatment initiation and linkage to care. The patients are determined to be responders by 90 days and therefore receive no active follow up.
  Interventions: Behavioral: SUN
- SUN followed by ED-ITT (Active Comparator): In Arm B, participants are randomized to receive SUN-assisted treatment initiation and linkage to care. The patients are determined to be non-responders within 90 days and are subsequently randomized into the ED-ITT condition to receive ongoing buprenorphine treatment by an ED-based interim treatment team.
  Interventions: Behavioral: SUN; Behavioral: ED-ITT
- SUN followed by ED-ITT + BHS (Active Comparator): In Arm C, participants are randomized to receive SUN-assisted treatment initiation and linkage to care. The patients are determined to be non-responders within 90 days and are subsequently randomized into the ED-ITT + BHS condition to receive ongoing buprenorphine treatment by an ED-based interim treatment team augmented with a behavioral health consultant who will provide behavioral health support for up to 3 months.
  Interventions: Behavioral: SUN; Behavioral: ED-ITT + BHS
- SUN + Telebridge with no follow up (Active Comparator): In Arm D, participants are randomized to receive SUN-assisted treatment initiation and linkage to care plus SUN-assisted immediate telehealth connection to an outpatient provider. The patients are determined to be responders by 90 days and therefore receive no active follow up.
  Interventions: Behavioral: SUN + Telebridge
- SUN + Telebridge followed by ED-ITT (Active Comparator): In Arm E, participants are randomized to receive SUN-assisted treatment initiation and linkage to care plus SUN-assisted immediate telehealth connection to an outpatient provider. The patients are determined to be non-responders within 90 days and are subsequently randomized into the ED-ITT condition to receive ongoing buprenorphine treatment by an ED-based interim treatment team.
  Interventions: Behavioral: SUN + Telebridge; Behavioral: ED-ITT
- SUN + Telebridge followed by ED-ITT + BHS (Active Comparator): In Arm F, participants are randomized to receive SUN-assisted treatment initiation and linkage to care plus SUN-assisted immediate telehealth connection to an outpatient provider. The patients are determined to be non-responders within 90 days and are subsequently randomized into the ED-ITT + BHS condition to receive ongoing buprenorphine treatment by an ED-based interim treatment team augmented with a behavioral health consultant who will provide behavioral health support for up to 3 months.
  Interventions: Behavioral: SUN + Telebridge; Behavioral: ED-ITT + BHS

INTERVENTIONS:
Behavioral: SUN — The SUN helps patients initiate buprenorphine treatment in the hospital, connects patients to follow-up care by facilitating appointments at outpatient clinics, addresses barriers to care, and serves as a resource for patients and clinicians. The SUN also advocates for a harm-reduction culture, models respectful interactions with people who use drugs and provides technical assistance to hospital staff to reduce stigma and discrimination.
  Arms: SUN followed by ED-ITT; SUN followed by ED-ITT + BHS; SUN with no follow up
Behavioral: SUN + Telebridge — TeleBridge consists of an immediate telehealth connection to a buprenorphine provider affiliated with the CA Bridge program who has expertise facilitating pharmacotherapy with individuals with OUD. TeleBridge addresses barriers to initiation of buprenorphine by reducing long wait times and the inability of the outpatient setting to initiate treatment on demand. TeleBridge also eliminates the need for patients to meet system-level requirements (e.g. on time for appointments during working hours while wearing appropriate attire) to obtain follow-up care. TeleBridge is a more resource-intensive form of care because it involves developing formalized relationships with outpatient providers and implementing telehealth protocols. TeleBridge is feasible based on the increased use of telehealth to expand post-ED care pathways.
  Arms: SUN + Telebridge followed by ED-ITT; SUN + Telebridge followed by ED-ITT + BHS; SUN + Telebridge with no follow up
Behavioral: ED-ITT — Enrolled patients who have not filled an outpatient buprenorphine (BUP) prescription at 30 days, return to the ED with an OUD-related event, or self-report nonadherence to the prescribed BUP are considered non-responders, and randomly assigned to a second stage intervention. For non-responders randomized to receive ongoing BUP treatment by an ED-based interim treatment team (ED-ITT), the SUN and Site PI (an ED physician with expertise in addiction medicine) will meet weekly to review the SUN's caseload, using a patient registry that has been modified for the trial. The registry: 1) prompts/documents proactive SUN outreach up to 3 additional months for non-responders, with an emphasis on prioritizing subsequent outreach to patients who have not yet engaged with outpatient care, or who are at risk of dropping out if the patient have transitioned; and 2) documents when the ED provider prescribes transitional BUP and when the patient would be due for a new prescription.
  Arms: SUN + Telebridge followed by ED-ITT; SUN followed by ED-ITT
Behavioral: ED-ITT + BHS — Enrolled patients who have not filled an outpatient buprenorphine (BUP) prescription at 30 days, return to the ED with an OUD-related event, or self-report to the SUN nonadherence to the prescribed BUP will be considered non-responders, and randomly assigned to a second stage intervention. For non-responders randomized to receive ongoing BUP treatment from the ED-ITT+BHS, Behavioral Health Support (BHS) will be added to ED-ITT and include a weekly caseload review with an externally-affiliated psychiatrist with expertise in addiction medicine who will make mental health and substance use treatment recommendations, both pharmacological and behavioral, to the ED provider and SUN for up to 3 months. The consultant may also ask the SUN to do a more detailed behavioral health assessment, if insufficient information is available to make treatment recommendations. All prescriptions will be written by the ED provider.
  Arms: SUN + Telebridge followed by ED-ITT + BHS; SUN followed by ED-ITT + BHS

SUMMARY:
The ADAPT-ED study is a two-stage, sequential multiple assignment randomized trial (SMART) to inform the development of an adaptive intervention that is optimally effective in increasing long-term buprenorphine use for adults presenting to the ED with probable opioid use disorder (OUD).

DETAILED DESCRIPTION:
The ADAPT-ED study is a two-stage, sequential multiple assignment randomized trial (SMART) to inform the development of an adaptive intervention that is optimally effective in increasing long-term buprenorphine use for adults presenting to the ED with probable OUD. The trial includes (1) two first stage components: the CA Bridge Model with Substance Use Navigator assisted treatment initiation and linkage to care (SUN) or CA Bridge plus immediate telehealth connection to an outpatient provider (SUN+TeleBridge); (2) a dynamic tailoring variable describing (non) response to the first stage: whether the patient has not filled an outpatient buprenorphine prescription at 30 days or whether the patient returns to the ED with an OUD-related event or self-reports non-adherence to buprenorphine within the first 90 days; (3) two second-stage components for non-responders; either ongoing buprenorphine treatment by an ED-based interim treatment team (ED-ITT) or ED-ITT augmented with behavioral health support (ED-ITT+BHS). First-stage responders will receive no further active intervention unless the participant returns to the ED or notifies the SUN about no longer taking buprenorphine within 90 days of study enrollment.

Hypothesis 1: The investigators hypothesize that the most intensive Adaptive Treatment Strategy (ATS) will lead to (a) more days of buprenorphine use and (b) a longer time to overdose, self-harm, or death compared to the least intensive ATS.

Hypothesis 2: The investigators hypothesize that (a) SUN+TeleBridge in the first stage of the ATS and (b) ED-ITT+BHS in the second stage of the ATS will each lead to more days of buprenorphine use and a longer time to overdose, self-harm, or death within the first 12 months compared to SUN and ED-ITT, respectively, and (c) there is a synergistic positive effect of receiving both SUN+TeleBridge and ED-ITT+BHS on days of buprenorphine use.

Hypothesis 3: The investigators hypothesize that the effect of SUN+TeleBridge versus SUN and the effect of ED-ITT+BHS versus ED-ITT among first stage non-responders will be larger among those with (a) a history of overdose at baseline and (b) co-occurring depression or PTSD at baseline relative to those who do not have either or those conditions.

ELIGIBILITY:
Inclusion Criteria:

* Presented for ED care at ARMC
* Age 18 or older
* Probable OUD diagnosis
* Speak and understand English or Spanish
* Have capacity to give informed consent
* Provide a signed and dated informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The number of days a buprenorphine prescription was filled in the 6 months after enrollment | 6 months from date of enrollment

SECONDARY OUTCOMES:
The time to a composite measure of overdose, suicide, self-harm and death | 6 months from date of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be destroyed in accordance with RAND Survey Research Group institutional policies (RAND SRG follows Federal guidelines, currently 7 years following study completion).